CLINICAL TRIAL: NCT00452855
Title: Postoperative Nausea and Vomiting Are Similar When Propofol or Sevoflurane Are Used as Adjuvant to Remifentanil During Anaesthesia for Gynaecological Surgery
Brief Title: Sevoflurane-Remifentanil Anaesthesia. The Risk of Post Operative Nausea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Jutland Regional Hospital (Other)
Collaborators: Nielsen, Jens OD, M.D. (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PropSevoRemi
Record Dates: First submitted 2007-03-26; First posted 2007-03-28 (Estimated); Last update posted 2007-03-29 (Estimated); Status verified 2007-03

CONDITIONS: Nausea; Vomiting
Keywords: Nausea; Vomiting; Post operative; Propofol remifentanil anaesthesia; Sevoflurane remifentanil anaesthesia
MeSH Terms: conditions — Nausea; Vomiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Sevoflurane-remifentanil anaesthesia

SUMMARY:
The purpose of this study is to determine whether sevoflurane-remifentanil anaesthesia is similar to propofol-remifentanil anaesthesia concerning post- operative nausea and vomiting.

DETAILED DESCRIPTION:
Propofol and sevoflurane anaesthesia are used world wide at the anaesthetists discretion.

Propofol is superior to inhalational anaesthetics as anaesthesia for patients at risk of post operative nausea and vomiting (PONV) as PONV is diminished. However, when remifentanil is used as adjuvant to sevoflurane, the total dose of the latter is reduced.

Therefore, we wanted to investigate if sevoflurane-remifentanil anaesthesia is similar to propofol-remifentanil anaesthesia with emphasis on nausea, vomiting and total PONV during 24 hours.

In the post anaesthesia care unit (PACU) and in the surgical ward nausea was scored on a visual analogue score. Vomiting was registered.

ELIGIBILITY:
Inclusion Criteria:

* Females younger than 50 years
* ASA I-II
* Scheduled to gynaecological laparotomies or laparoscopies

Exclusion Criteria:

* Medication known to act anti-emetic
* ASA status greater than II
* Malignant hyperthermia
* Allergy to the drugs used.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160
Dates: Start 2002-01; Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Nausea, incidence and intensity ( VAS score )in PACU and surgical ward
Vomiting, incidence in PACU and surgical ward
Total PONV after 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jens Ole Dich JO Nielsen, MD, Principal Investigator
Locations (1):
- Viborg Hospital, Viborg, Denmark